CLINICAL TRIAL: NCT07312084
Title: The Effect of Two Different Types of Hourglasses on Pain, Fear, and Anxiety During Blood Collection in Children: A Randomized Controlled Trial
Brief Title: The Effect of Two Different Types of Hourglasses on Pain, Fear, and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Demir Kösem, Associate Professor, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HakkariUO
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pain; Fear; Anxiety; Procedural Anxiety; Procedural Pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Liquid Gel-Based Hourglass Group: Children in this group will be administered a liquid gel-based hourglass as a non-pharmacological method. During blood collection, the hourglass will be kept in the children's view and, accompanied by the researcher or parent, will be turned, and the children will observe the flow of moving bubbles in the hourglass.
  Sand-Based Hourglass Group: Children in this group will be administered a conventional sand-based hourglass as a non-pharmacological method. During blood collection, the hourglass will be kept in the children's view and, accompanied by the researcher or parent, will be turned, and the children will observe the flow of sand grains.
  Control Group: Children in this group will not receive any pharmacological or non-pharmacological interventions other than routine blood collection.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to prevent bias, support will be obtained from an independent statistician. In addition, data will be collected by a nurse who does not know the groups not included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liquid Gel-Based Hourglass (Experimental): The liquid gel-based hourglass used in the study is approximately 13-14 cm long and made of high-quality plastic. It contains a highly viscous colored gel, which flows slowly and regularly in a drop-like pattern. These hourglasses are used during interventions not to measure time but to increase visual focus, distract attention, and provide a calming effect.
  Interventions: Other: Liquid Gel-Based Hourglass
- Sand-Based Hourglass (Experimental): The sand-based hourglass used in the study is approximately 8.5 cm long and made of durable plastic and glass. It contains colored, fine-grained, dry sand. It's a classic mechanism that relies on the fine-grained sand flowing from the upper chamber to the lower chamber under the influence of gravity. This type of hourglass is used as a helpful tool to distract children and reduce procedural anxiety during the intervention.
  Interventions: Other: Sand-Based Hourglass
- Control Group (No Intervention): Children in this group will not receive any pharmacological or non-pharmacological intervention other than routine blood collection.

INTERVENTIONS:
Other: Liquid Gel-Based Hourglass — The liquid gel-based hourglass used in the study is approximately 13-14 cm long and made of high-quality plastic. It contains a highly viscous colored gel, which flows slowly and regularly in a drop-like pattern. These hourglasses are used during interventions not to measure time but to increase visual focus, distract attention, and provide a calming effect.
  Arms: Liquid Gel-Based Hourglass
Other: Sand-Based Hourglass — The sand-based hourglass used in the study is approximately 8.5 cm long and made of durable plastic and glass. It contains colored, fine-grained, dry sand. It's a classic mechanism that relies on the fine-grained sand flowing from the upper chamber to the lower chamber under the influence of gravity. This type of hourglass is also used as a helpful tool to distract children and reduce procedural anxiety during the intervention.
  Arms: Sand-Based Hourglass

SUMMARY:
This research will be conducted as a pre-test-post-test parallel group randomized controlled experimental study to determine the effects of two different types of hourglasses (liquid gel-based hourglass and sand-based hourglass) used for distraction during blood collection in children aged 5-10 years on pain, fear, and anxiety and the comparative effectiveness of these methods.

Research Hypotheses H1: The mean pain, fear, and anxiety scores of children who used a liquid gel-based hourglass during blood collection were significantly lower than the mean scores of children in the control group.

H2: The mean pain, fear, and anxiety scores of children who used a sand-based hourglass during blood collection were significantly lower than the mean scores of children in the control group.

H3: The use of a liquid gel-based hourglass and a sand-based hourglass during blood collection had different effects on the mean pain, fear, and anxiety scores of children.

DETAILED DESCRIPTION:
Pain, fear, and anxiety experienced by children during medical procedures constitute a significant clinical and psychosocial concern. Venipuncture, particularly common among invasive procedures performed on children aged 5-10 years, can trigger strong emotional reactions in this age group. These reactions may negatively affect not only the procedure itself but also children's long-term trust in the healthcare system, treatment adherence, and tolerance of future procedures.

Failure to effectively manage the anxiety and fear that arise during invasive procedures in children may lead to movement, increased pain, delays in the procedure, and challenges in terms of staff safety. Moreover, children who experience high levels of fear and anxiety may later avoid similar procedures, which poses a serious risk for access to healthcare services and adherence to treatment. Therefore, identifying and optimizing non-pharmacological, low-cost, and feasible methods used during invasive procedures is of utmost importance.

One of the non-pharmacological strategies used to reduce pain, fear, and anxiety during invasive procedures in children is active and passive distraction. Active distraction methods involve the child's engagement in surrounding activities such as playing games, crafts and coloring, tablet/computer games, role-play, and storytelling. These methods require the child to use hand-eye coordination, cognitive skills, or imagination and often reduce pain and anxiety more effectively. Passive distraction methods rely on the child's observation or listening to an activity and include watching videos/cartoons, listening to music or stories, and observing visual toys (e.g., sand timers). These methods provide visual and auditory stimuli that help redirect attention away from painful cues and are generally easy to implement. In summary, while active methods involve the child's active participation in the process, passive methods rely solely on focusing on an external stimulus. Studies in the literature indicate that both methods play an important role in reducing pain, fear, and anxiety experienced by children during invasive procedures.

Among passive distraction methods, sand timers are used as visual toys. The reason for selecting two different types of sand timers for children is the potential for their visual and cognitive stimulus properties to influence levels of pain, fear, and anxiety differently. The traditional sand-based timer offers a simple visual stimulus by displaying the natural flow of sand and is familiar and calming for most children. In contrast, liquid gel-based timers provide a more dynamic and attention-grabbing stimulus through colorful liquid and varying flow speeds. These differing characteristics may influence how effectively children's attention can be diverted from painful cues during venipuncture. However, the literature on the effectiveness of visual distractors such as sand timers remains limited. Sand timers are simple, portable, and low-cost tools to capture children's attention, but differences between sand-based (traditional) and liquid gel-based versions-such as visual effects, flow speed, and color variations-have not been fully explored regarding their impact on pain, fear, and anxiety. This gap creates uncertainty about which type is more effective in clinical practice.

Systematically evaluating the effects of liquid gel-based and traditional sand timers on children's experience during invasive procedures may provide valuable evidence for nursing practice and pediatric care protocols. If simple and low-cost tools such as sand timers can reduce pain, fear, and anxiety during venipuncture, their widespread use may enhance children's procedural experiences and improve their cooperation and morale. Lower levels of pain and fear may help children move less during the procedure, increasing the safety of both the child and healthcare staff and supporting their compliance with future procedures. Furthermore, compared with medication- or device-based interventions, sand timers offer economic and logistical advantages; their ease of application in clinical settings and minimal training requirements make them highly feasible for practice.

This study aims to fill this gap in the literature, provide concrete recommendations regarding non-pharmacological support strategies for children during venipuncture, and contribute to improving children's healthcare experiences. It is also expected to support the efficient use of pediatric nurses' time and enhance the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Being between 5 and 10 years old,
* Agreeing to participate in the research by applying to the blood collection unit,
* Written consent being obtained from the parent,
* Physical and mental development being appropriate for the age.

Exclusion Criteria:

* Being outside the specified age range,
* Having a serious chronic disease or hematological disorder,
* Having developed serious trauma or intense anxiety due to a previous blood draw,
* Refusal to participate in the study or failure to obtain parental consent,
* Psychiatric or neurological disorders that may affect the implementation of the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain During Venous Blood Collection in Children (Wong-Baker Facial Pain Scale) | "1 year"
  "Pain is a specific unpleasant sensation originating from any part of the body, encompassing all past experiences of a person, whether or not due to an organic cause." The aim of the scale is to determine the level of pain based on numerical values corresponding to target facial expressions. Numerical values between 0 and 10 are used. A value of 0 indicates no pain, while a value of 10 indicates severe pain.
Fear During Venous Blood Collection in Children (Child Fear Scale) | "1 year"
  "It is a vital response that occurs as a response to a stimulus that is perceived as a specific pain or threat." The scale was developed to determine the level of fear in children aged 4-10 years. The scale uses facial expressions and is scored on a scale of "0-4". A score of "0" indicates no fear, while a score of "4" indicates excessive fear.
Anxiety During Venous Blood Collection in Children (Child Anxiety Scale - State) | "1 year"
  "It is a common psychological disorder that causes a person to have excessive and uncontrollable reactions to emotions such as worry, anxiety and fear." The CAS-D scale is shaped like a thermometer with a lightbulb at the bottom and horizontal lines at intervals going upwards. To measure CAS-D, the child is asked to indicate what they are feeling "right now." The scale is scored from 0 to 10. Children are asked to indicate their feelings of anxiety and nervousness from the bottom of the thermometer upwards (from least to most). Before using the scale, the child's sequencing skills are assessed. After being asked to count to ten, they are asked questions about which of two numbers is larger or smaller. Children who cannot follow the instructions or answer these questions are excluded from the scale.